CLINICAL TRIAL: NCT02365090
Title: Binocular iPad Sub-Study; Suppression in Amblyopia
Brief Title: Binocular iPad Sub-Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Retina Foundation of the Southwest (Other)
Responsible Party: Principal Investigator, Eileen Birch, Sr. Research Scientist, Retina Foundation of the Southwest
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Binocular iPad Sub-Study
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patching (occlusion therapy) (Active Comparator): 2 hours per day patching of the sound eye (for strabismic, anisometropic, and combined mechanism amblyopia) or current patching regimen (deprivation amblyopia)
  Interventions: Other: patching
- binocular games (Experimental): 1 hour per day (5 days per week) binocular game play
  Interventions: Other: binocular games

INTERVENTIONS:
Other: patching — covering the sound eye with a patch to force use of the amblyopic eye
  Other Names: occlusion therapy
  Arms: patching (occlusion therapy)
Other: binocular games — playing iPad games 1 hour per day 5 days per week to allow the child to use the amblyopic eye and the sound eye together
  Arms: binocular games

SUMMARY:
1. To determine whether a binocular iPad game app is effective in improving visual acuity and reducing interocular suppression in amblyopic children
2. To compare the amount of visual acuity improvement achieved with the binocular game app to the amount achieved with patching (standard treatment for amblyopia)

DETAILED DESCRIPTION:
Although patching treatment results in improved visual acuity for most amblyopic children, some fail to achieve normal visual acuity after months or years of treatment. Even among children who do achieve normal visual acuity with amblyopia treatment, the risk for recurrence of amblyopia is high. Patching treatment is based on the premise that amblyopia is a monocular disorder that can be treated by forcing use of the amblyopic eye. However, recent studies have elucidated a clear link between binocular dysfunction and the complex constellation of deficits that characterizes amblyopia, including visual acuity, vernier acuity, fixation instability, fusional suppression, and risk for residual and recurrent amblyopia. The association of binocular dysfunction and the myriad of monocular and binocular deficits in amblyopia has led us to hypothesize that amblyopia is a monocular consequence of a primary binocular obstacle to normal visual development.

Although binocular interaction does not normally occur in amblyopia, weak, noisy signals from the amblyopic eye can contribute to binocular vision if suppression by the fellow eye is reduced by signal attenuation, such as reduced stimulus contrast. In small cohorts of amblyopic adults and schoolchildren, repeated practice with a binocular Falling Blocks iPod game with reduced fellow eye contrast yielded modest visual acuity improvement after just 1-5 weeks (Hess et al 2010, 2012, 2014; Knox et al 2011; Li et al 2012). Recently, we showed that the same binocular game app approach(reduced fellow eye contrast) could be adapted for home use by amblyopic children on a larger iPad display (Li et al 2014; Birch et al 2014). These games also were effective in improving visual acuity, and the visual acuity gains were maintained for at least 6 months (Li et al 2014a, 2014b). The major limitation of both sets of studies was that the games were not very interesting and quickly became tedious to play day after day. To overcome this limitation, we propose to evaluate a new, more engaging binocular iPad adventure game to determine whether practice with a binocular iPad games app, with reduced fellow eye contrast, can improve visual acuity and reduce interocular suppression in children with amblyopia.One group of participants will include 56 children with anisometropic, strabismic, or combined mechanism amblyopia, age 4-10 years. The participants will be randomly assigned to patch 2 hours daily patching (standard-of-care treatment) or to play the iPad game app 1 hour per day 5 days per week for 2 weeks. Half of the children will have had no prior treatment for amblyopia and the other half will have had prior amblyopia treatment; these two subgroups will be randomized separately. A blocked randomization order will be provided in sealed envelopes by our consultant statistician. A second group of participants will include 40 children with deprivation amblyopia due to cataract. The participants will be randomly assigned to continue their patching regimen (if any) or to continue their current patching regimen and also play the iPad game app 1 hour per day 5 days per week for 4 weeks. iPads with the game app are loaned to the family for the duration of the study, Vision will be tested at baseline and at 2 weeks for the primary outcome of change in visual acuity (for strabismic, anisometropic, and combined mechanism amblyopia) or at baseline and 4 weeks (for deprivation amblyopia). At the primary outcome visit, the patching group will be crossed over to play the iPad game app 1 hour per day 5 days per week and return for a secondary outcome at 4 weeks (for strabismic, anisometropic, and combined mechanism amblyopia) or 8 weeks (for deprivation amblyopia). Families will have the option to discontinue or to continue with the game app for up to 8 weeks, with testing every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

Age 4-14 years Female and male Amblyopia with amblyopic eye visual acuity 20/40-20/125, fellow eye visual acuity 20/16-20/25, and interocular difference in visual acuity of 3 lines or more.

Anisometropic (with or without microtropia) or fully accommodative esotropia (no tropia present with glasses), or deprivation amblyopia Wearing glasses (if needed) for 8 weeks or no change in visual acuity with glasses wear for 4-6 weeks.

Must be able to demonstrate understanding and ability to play the Dig Rush game app during the enrollment visit.

Signed informed consent obtained

Exclusion Criteria:

Prematurity ≥8 weeks Coexisting ocular or systemic disease Developmental delay Poor ocular alignment (strabismus >5 prism diopters)

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2015-02; Primary Completion 2021-12-15 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity of the Amblyopic Eye HOTV (for children <7 y) or ETDRS for children 7+y | 2 weeks (for strabismic, anisometropic, and combined mechanism amblyopia); 4 weeks (for deprivation amblyopia)
  HOTV (for children <7 y) or ETDRS for children 7+y

SECONDARY OUTCOMES:
Visual Acuity of the Amblyopic Eye HOTV (for children <7 y) or ETDRS for children 7+y | 4 and 8 weeks (for strabismic, anisometropic, and combined mechanism amblyopia); 8 weeks (for deprivation amblyopia)
  HOTV (for children <7 y) or ETDRS for children 7+y
Stereoacuity Randot Preschool Stereoacuity Test | 2, 4, and 8 weeks (for strabismic, anisometropic, and combined mechanism amblyopia); 4 and 8 weeks (for deprivation amblyopia)
  Randot Preschool Stereoacuity Test
Interocular Suppression Dichoptic Motion Coherence Threshold (<7y) & Dichoptic Letter Contrast Threshold (7+ y) | 2, 4, and 8 weeks (for strabismic, anisometropic, and combined mechanism amblyopia); 4and 8 weeks (for deprivation amblyopia)
  Dichoptic Motion Coherence Threshold (<7y) & Dichoptic Letter Contrast Threshold (7+ y)
Fixation Stability BCEA during 30 sec fixation assessed using the EyeLink system | 2, 4, and 8 weeks (for strabismic, anisometropic, and combined mechanism amblyopia); 4 and 8 weeks (for deprivation amblyopia)
  BCEA during 30 sec fixation assessed using the EyeLink system

CONTACTS AND LOCATIONS:
Locations (1):
- Retina Foundation of the Southwest, Dallas, Texas, United States

REFERENCES:
- [Derived] Jost RM, Kelly KR, Birch EE. Risk of recurrence after cessation of dichoptic, binocular treatment of amblyopia. J AAPOS. 2023 Oct;27(5):298-300. doi: 10.1016/j.jaapos.2023.06.009. Epub 2023 Aug 23. PMID 37619861
- [Derived] Birch EE, Jost RM, Wang SX, Kelly KR. A pilot randomized trial of contrast-rebalanced binocular treatment for deprivation amblyopia. J AAPOS. 2020 Dec;24(6):344.e1-344.e5. doi: 10.1016/j.jaapos.2020.07.009. Epub 2020 Oct 16. PMID 33069871
- [Derived] Kelly KR, Jost RM, Dao L, Beauchamp CL, Leffler JN, Birch EE. Binocular iPad Game vs Patching for Treatment of Amblyopia in Children: A Randomized Clinical Trial. JAMA Ophthalmol. 2016 Dec 1;134(12):1402-1408. doi: 10.1001/jamaophthalmol.2016.4224. PMID 27832248

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-25): https://cdn.clinicaltrials.gov/large-docs/90/NCT02365090/Prot_SAP_000.pdf